CLINICAL TRIAL: NCT02588950
Title: Comparative Pharmacokinetics and Pharmacodynamics of Human Regular U-500 Insulin Administered Subcutaneously as a Bolus Via Syringe Versus Continuous Subcutaneous Insulin Infusion and Characterization of TID and BID Dosing at Steady State in High-Dose Insulin-Treated Subjects With Type 2 Diabetes Mellitus
Brief Title: A Study of U-500 Insulin (LY041001) in Participants With Type 2 Diabetes
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Slow enrollment
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 16021; B5K-EW-IBHG (Other: Eli Lilly and Company)
Record Dates: First submitted 2015-10-27; First posted 2015-10-28 (Estimated); Results first posted 2023-10-18 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Insulin, Regular, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Part A: U-500R Single Injection (Experimental): Bolus of U-500R administered via single subcutaneous (SC) injection.
  Interventions: Drug: U-500R
- Part A: U-500R CSII (Experimental): Bolus of U-500R administered via continuous subcutaneous insulin infusion (CSII).
  Interventions: Drug: U-500R
- Part B: U-500R TID (Experimental): U-500R administered thrice-daily (TID) via SC injection under steady state conditions for 5 to 10 days
  Interventions: Drug: U-500R
- Part B: U-500R BID (Experimental): U-500R administered twice-daily (BID) via SC injection under steady state conditions for 5 to 10 days
  Interventions: Drug: U-500R

INTERVENTIONS:
Drug: U-500R
  Other Names: Humulin R U-500; LY041001; Humulin

SUMMARY:
The purpose of this two-part study is to measure how much of the study drug gets into the blood stream and how long it takes the body to get rid of it. In Part A, each participant will receive two treatments, a single dose and a single dose with continuous infusion of U-500R insulin, both administered just under the skin. Participants who complete Part A will continue into Part B where they will be assigned to 1 of 2 treatments with U-500R insulin, injected either twice or three times daily under the skin for 5-10 days. This study can last from 7-14 weeks including initial screening and follow up.

ELIGIBILITY:
Inclusion Criteria:

* Males or females with type 2 diabetes mellitus (T2DM)
* Are current users of U-100, U-200 and/or U-300 insulin/analog as, basal, premixed and/or basal/bolus delivered with any injection device (pens and/or syringe/vial but excluding continuous subcutaneous infusion (CSII)/insulin pump use in the preceding 3 months), taking a total daily dose (TDD) of greater than or equal to (≥) 150 units (U) or at least one dose greater than (>) 100 U as part of a multiple daily injection (MDI) regimen and TDD less than or equal to (≤)3.0 units per kilogram (U/kg)
* Concomitant antihyperglycemic agent(s) (AHA) therapy may include: metformin (MET), dipeptidyl peptidase 4 inhibitors, pioglitazone (doses ≤30 milligrams per day (mg/day)), glucagon like peptide (GLP)-1 receptor agonists, sodium-glucose co-transporter-2 (SGLT2) inhibitors, except in combination with GLP-1 receptor agonists
* Participant's antihyperglycemic agent (AHA) therapy must have been stable for ≥3 months (except for weekly GLP-1 receptor agonists which must have been stable for ≥4 months)
* Have hemoglobin A1c (HbA1c) 7.5-11.5 percent (%)

Exclusion Criteria:

* Have type 1 diabetes mellitus (T1DM), or other types of diabetes mellitus apart from T2DM
* Have known hypersensitivities or allergies to insulin, excipients contained in insulin products, or related compounds
* Have used U-500R within 3 months prior to screening
* Have used rosiglitazone, pramlintide, once weekly or twice daily exenatide, or other injectable or oral antihyperglycemic agent(s) not listed in the inclusion criterion; or are taking oral antidiabetic medications at doses exceeding the respective product labels
* Have had a blood transfusion or severe blood loss within 3 months prior to screening or have known hemoglobinopathy, hemolytic anemia, or sickle cell anemia which may affect reliability of HbA1c measurements

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2016-01-12 (Actual); Primary Completion 2017-05-25 (Actual); Study Completion 2017-05-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- Profil Institute for Clinical Research, Chula Vista, California, United States

REFERENCES:
- See also: Click here for more information about this study: A Study of U-500 Insulin (Humulin LY041001) in Participants With Type 2 Diabetes — http://www.lillytrialguide.com/en-US/studies/type-2%20diabetes/IBHG#?postal=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Two parts study with Part A (Periods 1 & 2) & Part B (Period 3). Part A:Participants received study drug either by subcutaneous(SC) or continuous subcutaneous insulin infusion (CSII) as per the dosing sequence.
  Part B: Participants received study drug via SC injection either twice daily (BID) or three times daily (TID) as per the dosing sequence.
Groups:
- Sequence 1: Participants received 100- Unit (U) of human regular U-500 insulin (U-500R) by subcutaneous (SC) injection in period 1 and 4.25 U/hour U-500R basal infusion for 12 hours prior to and during the 24 hour clamp plus a 100-U of U-500R via continuous SC insulin infusion (CSII) in period 2 and U-500R administered thrice daily via SC injection in period 3.
- Sequence 2: Participants received 4.25 U/hour U-500R basal infusion for 12 hours prior to and during the 24 hour clamp plus a 100-U of U-500R via continuous SC insulin infusion (CSII) in period 1 and 100-U of human regular U-500 insulin (U-500R) by subcutaneous (SC) injection in period 2 and U-500R administered twice daily via SC injection in period 3.
- Sequence 3: Participants received 100-U of human regular U-500 insulin (U-500R) by subcutaneous (SC) injection in period 1 and 4.25 U/hour U-500R basal infusion for 12 hours prior to and during the 24 hour clamp plus a 100-U of U-500R via continuous SC insulin infusion (CSII) in period 2 and U-500R administered twice daily via SC injection in period 3.
- Sequence 4: Participants received 4.25 U/hour U-500R basal infusion for 12 hours prior to and during the 24 hour clamp plus a 100-U of U-500R via continuous SC insulin infusion (CSII) in period 1 and 100-U of human regular U-500 insulin (U-500R) by subcutaneous (SC) injection in period 2 and U-500R administered thrice daily via SC injection in period 3.
Period: Period 1 (Part A)
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4
Started | 3 | 2 | 3 | 3
Received at Least One Dose of Study Drug | 3 | 2 | 3 | 3
Completed | 3 | 2 | 3 | 3
Not Completed | 0 | 0 | 0 | 0
Period: Period 2 (Part A)
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4
Started | 3 | 2 | 3 | 3
Completed | 3 | 2 | 2 | 3
Not Completed | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0
Period: Period 3 (Part B)
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4
Started | 3 | 2 | 2 | 3
Completed | 3 | 2 | 2 | 2
Not Completed | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- Overall: Participants received 100-U of human regular U-500 insulin (U-500R) by subcutaneous (SC) injection or 4.25 U/hour U-500R basal infusion for 12 hours prior to and during the 24 hour clamp plus a 100-U of U-500R via continuous SC insulin infusion (CSII) in Part A (periods 1 & 2), and U-500R administered twice or thrice daily via SC injection in part B (period 3) as per the dosing sequence in each period.
Arm/Group | Overall
Number analyzed (Participants) | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.2 (7.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 7
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 6
  More than one race | 1
  Unknown or Not Reported | 0
Body mass index [Mean (Standard Deviation); unit: Kilogram per square meter (kg/m^2)] | 39.63 (8.59)

OUTCOME MEASURES:

1. Primary Outcome: Part A: Pharmacokinetics (PK): Time to Maximum Drug Concentration (Tmax) of U-500R
Description: Part A: Pharmacokinetics (PK): Time to Maximum Drug Concentration (Tmax) of U-500R.
Time Frame: Period 1 and 2: -0.5, 0, 0.5, 1, 2, 3, 4, 6, 7, 8, 12, 16, 24 hours (h) post dose
Population: All randomized participants who received at least one dose of study drug and had evaluable PK data in part A.
Measure: Median (Full Range); unit: Hours (h)
Groups:
- 100-U Bolus U-500R SC: Participants received 100-U of human regular U-500 insulin (U-500R) by subcutaneous (SC) injection.
- 100-U Bolus U-500R CSII: Participants received 4.25 U/hour U-500R basal infusion for 12 hours prior to and during the 24 hour clamp plus a 100-U of U-500R via continuous SC insulin infusion (CSII).
Arm/Group | 100-U Bolus U-500R SC | 100-U Bolus U-500R CSII
Number analyzed (Participants) | 11 | 11
Hours (h) | 6 [0.5 to 8] | 5 [0.5 to 12]
Statistical Analysis 1: Comparison: 100-U Bolus U-500R SC vs 100-U Bolus U-500R CSII; Test type: Superiority; Mixed Models Analysis; Geometric LSMean Ratio = 1.46, 90% CI 2-sided [1.08 to 1.97]

2. Primary Outcome: Part B: Pharmacokinetics: Area Under the Concentration Versus Time Curve From Zero to 24 Hours Postdose (AUC[0-24]) of U-500R
Description: Part B: Pharmacokinetics: Area Under the Concentration Versus Time Curve from Zero to 24 Hours Postdose (AUC[0-24]) of U-500R.
Time Frame: Period 3: -0.5, 0, 0.5, 1, 2, 3, 4, 5, 6, 7, 9, 11, 12, 13, 15, 18, 24h post dose
Population: All randomized participants who received at least one dose of study drug and had evaluable PK data in part B.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Picomoles hour per liter (pmol*h/L)
Groups:
- U-500R BID: Participants received U-500R twice daily by SC injection for 5 to 10 days.
- U-500R TID: Participants received U-500R thrice daily by SC injection for 5 to 10 days.
Arm/Group | U-500R BID | U-500R TID
Number analyzed (Participants) | 3 | 5
Picomoles hour per liter (pmol*h/L) | 7790 (57) | 11700 (77)

3. Primary Outcome: Part B: Pharmacokinetics: Maximum Observed Drug Concentration (Cmax) of U-500R
Description: Pharmacokinetics: Maximum Observed Drug Concentration (Cmax) of U-500R.
Time Frame: Period 3: -0.5, 0, 0.5, 1, 2, 3, 4, 5, 6, 7, 9, 11, 12, 13, 15, 18, 24h post dose
Population: All randomized participants who received at least one dose of study drug and had evaluable PK data in part B.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Pico mole per liter (Pmol/L)
Arm/Group | U-500R BID | U-500R TID
Number analyzed (Participants) | 4 | 5
Pico mole per liter (Pmol/L) | 699 (47) | 1050 (82)

4. Primary Outcome: Part B: Pharmacodynamics: Maximum Glucose Infusion Rate (Rmax) of U-500R
Description: Pharmacodynamics: Maximum Glucose Infusion Rate (Rmax) of U-500R.
Time Frame: Period 3 day 1: 0, 0.5, 1, 2, 3, 4, 5, 6, 7, 9, 11, 12, 13, 15, 18h post dose
Population: All randomized participants who received at least one dose of study drug and had evaluable PK data in part B.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Milligram per Minute (mg/min)
Arm/Group | U-500R BID | U-500R TID
Number analyzed (Participants) | 4 | 5
Milligram per Minute (mg/min) | 524 (30) | 588 (28)

5. Secondary Outcome: Part A: Pharmacokinetics: Area Under The Concentration Versus Time Curve From Time Zero to Last Time Point With A Measurable Concentration (AUC[0-tlast]) of U-500R
Description: Part A: Pharmacokinetics: Area Under The Concentration Versus Time Curve From Time Zero to Last Time Point With A Measurable Concentration (AUC[0-tlast]) of U-500R.
Time Frame: Period 1 and 2: -0.5, 0, 0.5, 1, 2, 3, 4, 6, 7, 8, 12, 16, 24h post dose
Population: All randomized participants who received at least one dose of study drug and had evaluable PK data in Part A.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Picomole hours per liter (pmol^h/L)
Arm/Group | 100-U Bolus U-500R SC | 100-U Bolus U-500R CSII
Number analyzed (Participants) | 11 | 11
Picomole hours per liter (pmol^h/L) | 5230 (35) | 6070 (70)
Statistical Analysis 1: Comparison: 100-U Bolus U-500R SC vs 100-U Bolus U-500R CSII; Test type: Superiority; Mixed Models Analysis; Geometric LSMean Ratio = 0.885, 90% CI 2-sided [0.761 to 1.03]

6. Secondary Outcome: Part A: Pharmacodynamics (PD): Time to Rmax (tRmax) of U-500R
Description: Part A: Pharmacodynamics (PD): Time to Rmax (tRmax) of U-500R.
Time Frame: Period 1 and 2: 0, 0.5, 1, 2, 3, 4, 6, 7, 8, 12, 16, 24h post dose
Population: All randomized participants who received at least one dose of study drug and had evaluable PD data in Part A.
Measure: Geometric Least Squares Mean (Geometric Coefficient of Variation); unit: Hour (h)
Arm/Group | 100-U Bolus U-500R SC | 100-U Bolus U-500R CSII
Number analyzed (Participants) | 11 | 11
Hour (h) | 8.50 (31) | 8.53 (35)
Statistical Analysis 1: Comparison: 100-U Bolus U-500R SC vs 100-U Bolus U-500R CSII; Test type: Superiority; Median Difference (Final Values) = 0.900, 90% CI 2-sided [-1.60 to 2.60]

7. Secondary Outcome: Part B: Pharmacokinetics: Time to Maximum Concentration (Tmax) of U-500R
Description: Part B: Pharmacokinetics: Time to Maximum Concentration (Tmax) of U-500R.
Time Frame: Period 3: -0.5, 0, 0.5, 1, 2, 3, 4, 5, 6, 7, 9, 11, 12, 13, 15, 18, 24h post dose
Population: All randomized participants who received at least one dose of study drug and had evaluable PK data in part B.
Measure: Median (Full Range); unit: Hours
Arm/Group | U-500R BID | U-500R TID
Number analyzed (Participants) | 4 | 5
Hours | 15 [5 to 18] | 15 [7 to 15]

8. Secondary Outcome: Part B: Pharmacodynamics: Total Amount of Glucose Infused (Gtot) of U-500R
Description: Pharmacodynamics: Total Amount of Glucose Infused (Gtot) of U-500R.
Time Frame: Period 3: 0, 0.5, 1, 2, 3, 4, 5, 6, 7, 9, 11, 12, 13, 15, 18, 24h post dose
Population: All randomized participants who received at least one dose of study drug and had evaluable PK data in part B.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Grams (g)
Arm/Group | U-500R BID | U-500R TID
Number analyzed (Participants) | 4 | 5
Grams (g) | 441 (27) | 510 (28)

9. Secondary Outcome: Part B: Pharmacodynamics: Time to Rmax (tRmax) of U-500R
Description: Part B: Pharmacodynamics: Time to Rmax (tRmax) of U-500R.
Time Frame: Period 3: 0, 0.5, 1, 2, 3, 4, 5, 6, 7, 9, 11, 12, 13, 15, 18, 24h post dose
Population: All randomized participants who received at least one dose of study drug and had evaluable PD data in part B.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | U-500R BID | U-500R TID
Number analyzed (Participants) | 4 | 5
Hours | 12.4 (64) | 13.8 (7)

ADVERSE EVENTS:
Time Frame: Up to 72 weeks
Arm/Group | 100-U Bolus U-500R SC | 100-U Bolus U-500R CSII | U-500R BID | U-500R TID
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/11 | 0/4 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/11 | 0/4 | 0/6
Other Adverse Events (participants affected / at risk) | 4/11 | 3/11 | 2/4 | 2/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 100-U Bolus U-500R SC (N=11) | 100-U Bolus U-500R CSII (N=11) | U-500R BID (N=4) | U-500R TID (N=6)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal disorder (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infusion site extravasation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Medical device site swelling (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peripheral swelling (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Procedural complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Increased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Priapism (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Petechiae (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eye laser surgery (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on PI is that sponsor can review results communications and comment 30 days prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 60 days. If PI is unwilling to delay the results communication then PI can remove the information that sponsor has specified it reasonably believes would jeopardize its intellectual property interests.

DOCUMENTS (2):
  • Study Protocol (2016-06-07): https://cdn.clinicaltrials.gov/large-docs/50/NCT02588950/Prot_000.pdf
  • Statistical Analysis Plan (2015-09-21): https://cdn.clinicaltrials.gov/large-docs/50/NCT02588950/SAP_001.pdf